CLINICAL TRIAL: NCT04020588
Title: Effect of Anti-inflammatory Treatments on the Symptoms, Cognition, and Functioning of Adolescents With Schizophrenia
Brief Title: Anti-inflammatories and Adolescent Schizophrenia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Psiquiatrico Infantil Dr. Juan N. Navarro, Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: II3/02/0618
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Schizophrenia
Keywords: schizophrenia; adolescents; inflammation; anti-inflammatory
MeSH Terms: conditions — Schizophrenia; Inflammation | interventions — Celecoxib; Minocycline

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Celecoxib (Active Comparator): Celecoxib 200 mg twice a day
  Interventions: Drug: Celecoxib 200mg
- Minocycline (Active Comparator): Minocycline 100 mg twice a day
  Interventions: Drug: Minocycline 100mg
- Placebo (Placebo Comparator): Placebo capsules twice a day
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Celecoxib 200mg — Will be administered for 6 weeks
  Other Names: Minocycline 100 mg; Minocycline
  Arms: Celecoxib
Drug: Placebo oral capsule — Will be administered for 6 weeks
  Other Names: Placebo
  Arms: Placebo
Drug: Minocycline 100mg — Will be administered for 6 weeks
  Other Names: Minocycline
  Arms: Minocycline

SUMMARY:
A double-blind controlled trial assessing the efficacy of anti-inflammatories on symptoms and cognition of adolescents with schizophrenia

DETAILED DESCRIPTION:
Patients will be evaluated to confirm the diagnosis of schizophrenia, duration of the disease and record a history of atopic diseases or recurrent infections throughout life. The PANSS, PSP, and MCCB battery scales will be administered. A blood sample will be taken for the determination of markers of inflammation before the start of pharmacological treatment.

Patients will start the antipsychotic medication assigned by their treating physician. They will also be assigned randomly to the treatment arm. The study drug will be provided by the research team under the presentation of capsules containing Celecoxib 200 mg, Minocycline 100 mg or Placebo, and patients will be instructed to take one capsule every 12 hrs daily.

The patient will be reassessed with PANSS, PSP, and MCCB after completing 6 weeks of pharmacological treatment, type and dose of medication will be recorded and serum markers of inflammation will be determined again.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizophreniform disorder.
* Patients in their first psychotic episode or previously diagnosed
* No specific pharmacological treatment (antipsychotic at therapeutic doses in regular doses) in the previous two weeks.
* Have a responsible parent or guardian.

Exclusion Criteria:

* Active infection

  * Chronic somatic diseases, including autoimmune diseases
  * Comorbidity with anorexia, substance use disorders
  * Pregnancy
  * Use of anti-inflammatory medications or antibiotics

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2019-02-25 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Symptom severity: Positive and Negative Syndrome Scale score | six weeks
  Change in the Positive and Negative Syndrome Scale score, which comprises 33 items which can be scored from 1 (absent) to 7 (extreme), evaluating an array of symptoms including positive, negative, neuromotor, depressive and anxious, and involves the use of data from patient reports, caregiver reports, and clinical observations. The total score is the sum or all the items, the maximum score is 231. The higher values represent a worse outcome
Cognition: MATRICS Consensus Cognitive Battery (MCCB) scores | six weeks
  Change in MCCB scores. The MCCB is comprised of 9 tests that reflect 7 dimensions of neurocognitive dysfunction in schizophrenia, including: Speed of Processing, Attention/Vigilance, Working Memory, Verbal Learning, Visual Learning, and Reasoning and Problem Solving and Social Cognition. The MCCB scoring program yields the domain scores and a composite score which are standardized to the same T-score measurement scale with a mean of 50 and an SD of 10 based upon the normative data.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Psiquiatrico Infantil, Mexico City, Ni Ee.uu. Ni Canadá, Mexico

IPD SHARING:
Plan to Share IPD: No